CLINICAL TRIAL: NCT00878904
Title: A Phase I Trial of Panobinostat (LBH589) and Epirubicin in Patients With Solid Tumor Malignancies
Brief Title: Panobinostat and Epirubicin in Treating Patients With Metastatic Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000639080; UCSF-09991; NOVARTIS-CLBH589C
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Epirubicin; Panobinostat; Gene Expression Profiling; Blotting, Western; Immunologic Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment with Panobinostat and Epirubicin (Experimental)
  Interventions: Drug: epirubicin hydrochloride; Drug: panobinostat; Genetic: gene expression analysis; Genetic: protein expression analysis; Genetic: western blotting; Other: immunologic technique; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: panobinostat
Genetic: gene expression analysis
Genetic: protein expression analysis
Genetic: western blotting
Other: immunologic technique
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Panobinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as epirubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving panobinostat together with epirubicin may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of panobinostat when given together with epirubicin in treating patients with metastatic malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety, tolerability, maximum tolerated dose (MTD), and recommended phase II dose of panobinostat when administered with epirubicin hydrochloride in patients with metastatic malignant solid tumors.

Secondary

* To determine the correlation between the pharmacokinetic profile of panobinostat drug levels and the pharmacodynamic effect of panobinostat on histone acetylation in peripheral blood mononuclear cells (PBMCs).
* To determine the effect of panobinostat on histone acetylation and chromatin remodeling proteins (HP-1, DNMT-1, SMC1-5, Topo II).
* To determine the relevance of HDAC1, HDAC2, HDAC3, and HDAC6 expression in PBMCs as a pharmacological marker and in biopsied tumors as a predictive marker for response in patients treated at the MTD.
* To document any objective response in these patients.

OUTLINE: This is a dose-escalation study of panobinostat.

Patients receive oral panobinostat on days 1, 3, and 5 and epirubicin hydrochloride IV on day 5. Treatment repeats every 21 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection at baseline and periodically during course 1 for panobinostat pharmacokinetic studies. Patients enrolled in the dose expansion cohort also undergo collection of tumor tissue samples by fine needle aspiration at baseline and on day 5 of course 1 (after panobinostat infusion). Blood and tissue samples are analyzed for histone acetylation, chromatin remodeling genes and proteins (HP-1, DNMT-1, SMC1-5, Topo II), and HDAC enzyme expression by immunofluorescence and western blotting.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed solid tumor malignancy for which no curative therapy exists

  * Metastatic disease
* Measurable or evaluable disease (i.e., elevated CA-125 or elevated PSA for patients with ovarian cancer or prostate cancer, respectively)
* Disease amenable to biopsy AND patient willing to undergo biopsies (for patients enrolled in the dose expansion cohort only)
* No uncontrolled CNS metastasis

  * Stable CNS metastasis allowed provided patient has undergone complete surgical resection, gamma knife radiotherapy (for isolated lesions) or whole-brain radiotherapy AND the metastasis has been stable for ≥ 6 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC > 3,000/mm³
* ANC > 1,500/mm³
* Hemoglobin > 9.0 g/dL (RBC transfusion allowed)
* Platelet count > 100,000/mm³
* AST/ALT ≤ 1.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.3 times ULN
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min by 24-hour urine collection
* Total serum calcium (corrected for serum albumin) or ionized calcium ≥ lower limit of normal
* Serum potassium ≥ 4.0 mEq/L (supplementation allowed)
* Serum magnesium normal (supplementation allowed)
* Serum sodium ≥ 130 mEq/L
* Serum albumin ≥ 3 g/dL
* Elevated alkaline phosphatase or gamma-glutamyl-transferase due to bone metastasis or liver metastasis allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method (including barrier) contraception during and for 3 months after completion of study treatment
* QTc < 460 ms
* No evidence of significant active infection (e.g., pneumonia, cellulitis, or wound abscess)
* No impaired cardiac function, including any of the following:

  * Complete left bundle branch block or use of a permanent cardiac pacemaker
  * Congenital long QT syndrome
  * History or presence of ventricular tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * QTcF > 470 msec on screening ECG
  * Right bundle branch block plus left anterior hemiblock (bifascicular block)
  * Atrial fibrillation (ventricular heart rate > 100 beats per minute)
  * Angina pectoris or acute myocardial infarction within the past 6 months
  * New York Heart Association class III-IV congestive heart failure
  * LVEF < 50% on baseline MUGA or ECHO
* No history of seizures

PRIOR CONCURRENT THERAPY:

* No prior cumulative anthracycline dose > 300 mg/m² of doxorubicin hydrochloride or > 480 mg/m² of epirubicin hydrochloride
* More than 5 days since prior valproic acid
* More than 3 weeks since prior and no other concurrent chemotherapy, hormonal therapy, radiotherapy, or experimental anticancer therapy for the primary disease
* No other concurrent HDAC inhibitors
* No concurrent medications that may induce torsades de pointes or cause QTc prolongation
* No other concurrent investigational or anticancer therapy
* No concurrent CYP3A4 inhibitors (including grapefruit or grapefruit juice) and/or CYP3A4 inducers
* No concurrent anti-arrhythmic therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09-13 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
Response as assessed by RECIST criteria | 30 post end of study drug estimated to be ~24 weeks
Progression as assessed by RECIST criteria | 30 post end of study drug estimated to be ~24 weeks
Adverse events and other symptoms as assessed by NCI CTCAE v3.0 | 30 post end of study drug estimated to be ~24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pamela N. Munster, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Derived] Thomas S, Aggarwal R, Jahan T, Ryan C, Troung T, Cripps AM, Raha P, Thurn KT, Chen S, Grabowsky JA, Park J, Hwang J, Daud A, Munster PN. A phase I trial of panobinostat and epirubicin in solid tumors with a dose expansion in patients with sarcoma. Ann Oncol. 2016 May;27(5):947-52. doi: 10.1093/annonc/mdw044. Epub 2016 Feb 21. PMID 26903311